CLINICAL TRIAL: NCT01588834
Title: Pilot Study to Examine Histological Characteristics of Mammographic Density With Molecular Breast Imaging: Part 2 - Premenopausal Women
Brief Title: Histology of Functional Density in Premenopausal Breast
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie Hruska, Principal Investigator, Mayo Clinic
Other Study IDs: 12-000458
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Dense Breasts; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — core biopsy samples from mammographically dense breast tissue
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: breast biopsy — ultrasound-guided core needle biopsy of healthy, mammographically dense breast tissue

SUMMARY:
The investigators hypothesize that knowledge of the functional behavior of areas of mammographic density will enable more specific identification of dense tissue at-risk for breast cancer, ultimately providing predictive information on an individual's risk of developing breast cancer.

DETAILED DESCRIPTION:
The specific aims are:

* In women with increased mammographic density (MD), determine the histological characteristics of functionally dense tissue compared to that of non-functionally dense tissue via core-needle biopsy of the breast.
* In women with increased mammographic density (MD), determine the correlations between the total percent area of functional density (FD) on MBI, percent density of MD on mammogram, and histological characteristics of dense tissue

ELIGIBILITY:
Inclusion Criteria:

* Ages 40 - 55 years
* Considered premenopausal or peri-menopausal
* Screening mammogram performed at Mayo Clinic Rochester within one year prior to the current MBI study which demonstrates
* Negative/benign assessment (BIRADS category 1-2) or Additional imaging recommended (BIRADS category 0), where the subsequent diagnostic workup results in a final negative/benign assessment (BIRADS category 1-2).
* No proliferative benign lesions (e.g. fibroadenomas) identified
* Heterogeneously dense or extremely dense parenchyma (BIRADs density category 3 or 4)
* MBI performed less than 3 days prior to biopsy demonstrating either marked FD or photopenic FD in an area of mammographically dense tissue amenable to biopsy.
* No use of exogenous hormonal drugs (e.g. hormonal contraceptives or sex steroid hormones) within six months prior to study biopsy
* Negative pregnancy test or surgically sterilized (for patients in whom a study MBI will be performed)

Exclusion criteria:

* Using any estrogen receptor modulating drugs (e.g., tamoxifen, raloxifene) or any aromatase inhibitors within six months prior to study biopsy.
* Prior diagnosis of bilateral breast cancer.
* Diagnosis of breast cancer in either breast within 3 years prior to study MBI.
* Diagnosis of any cancer, except breast cancer (see #3) or non-melanomatous skin cancer, for which patient has not been disease free for at least 5 years.
* Current breast symptoms
* Breast implants
* Known allergy to local anesthetic.
* History of bleeding complications from prior interventions
* Current use of anticoagulants (e.g., Coumadin or other blood thinners)
* Major medical condition

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with mammographically dense breasts who demonstrate either photopenic or marked background parenchymal uptake on MBI
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
proportion of epithelium vs stroma | within 3 days of functional density assessment on MBI

SECONDARY OUTCOMES:
Degree of lobular involution | within 3 days of functional density assessment on MBI
  Degree of lobular involution as assessed through qualitative and quantitative measurements will be compared between dense tissue which appears photopenic on MBI and dense tissue which appears functionally active on MBI.
Ki-67 cellular proliferation index | within 3 days of functional density assessment on MBI
  Degree of cellular proliferation as assessed through Ki-67 index will be compared between dense tissue which appears photopenic on MBI and dense tissue which appears functionally active on MBI.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie B Hruska, PhD R-D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bardwell Speltz L, Ghosh K, Visscher DW, Scott CG, Cole KC, Kroneman TN, Maxwell RW, Conners AL, Hunt KN, Rhodes DJ, Vachon CM, Hruska CB. Histologic correlates of background parenchymal uptake on molecular breast imaging. Breast Cancer Res. 2025 Dec 16;27(1):216. doi: 10.1186/s13058-025-02171-x. PMID 41402965
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0